CLINICAL TRIAL: NCT00367952
Title: An Open Label Long Term Safety Extension Study of Apricitabine in Treatment-experienced HIV-1 Infected Subjects
Brief Title: A Long Term, Safety Study of Apricitabine in HIV-infected Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avexa (Industry)
Responsible Party: Susan Cox, Avexa
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVX-201E
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infection
Keywords: HIV; apricitabine; drug resistance; reverse transcriptase; lamivudine
MeSH Terms: conditions — HIV Infections | interventions — apricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ATC 800mg BID (Experimental): 800mg ATC BID
  Interventions: Drug: apricitabine

INTERVENTIONS:
Drug: apricitabine — 800mg apricitabine twice daily orally for 96 weeks

SUMMARY:
The study will examine how safe and effective apricitabine is when given long term (as ongoing treatment) to HIV patients who have already completed the AVX-201 trial

DETAILED DESCRIPTION:
An ongoing study (AVX-201) is examining the safety and efficacy of apricitabine compared to 3TC in HIV patients who are failing therapy containing 3TC and have the presence of the M184V mutation in reverse transcriptase. This extension study (AVX-201E) is available to patients who complete the AVX-201 protocol.

Patients will continue to receive apricitabine open label for a further 96 weeks (making a total of 144 weeks from starting AVX-201) in addition to an optimised background. Safety markers and efficacy markers will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Completed AVX-201 protocol, Plasma HIV RNA <5000 copies/ml, CD4 cells >50

Exclusion Criteria:

* Pregnant or breastfeeding females, withdrawal from AVX-201

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Time to virological failure (DHSS definition) | week 144
incidence of AEs and laboratory abnormalities | Week 144
time to withdrawal due to AEs | Week 144

SECONDARY OUTCOMES:
Change from baseline HIV RNA | weeks 72, 96, 120, and 144
Proportion of subjects with plasma HIV RNA <400 and <50 copies/ml | at weeks 72, 96, 120, and 144
Change from baseline and change in ratio of CD4+ and CD8+ counts | at weeks 72, 96, 120, and 144

CONTACTS AND LOCATIONS:
Overall Officials: Susan W Cox, Ph D, Study Director — Avexa
Locations (1):
- Avexa (co-ordinating sites in Australia and Argentina), Melbourne, Victoria, Australia